CLINICAL TRIAL: NCT03969745
Title: Effects of Two-weeks of Time Restricted Feeding on Basal and Postprandial Metabolism in Healthy Men
Acronym: TRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-1705
Record Dates: First submitted 2019-04-30; First posted 2019-05-31 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Health
Keywords: chrononutrition; metabolism; body composition
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: All participants monitored for a one week baseline period before being allocated to either a caloric deficit group or a time-restricted feeding group for two weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted feeding (TRF) (Experimental): Participants restricted their daily energy intake window to between 8 am and 4 pm for two weeks. They were encouraged to not alter the quantity and composition of their diet or alter physical activity patterns.
  Interventions: Behavioral: Time restricted feeding
- Caloric deficit (Active Comparator): The investigators observed significant weight loss in the TRF group with participants reporting to consume ~400 kilocalories less per day. Therefore the investigators added a caloric deficit group to control for the effects of weight loss on metabolism. Total energy expenditure was measured for one week and was used to prescribe a 400 kilocalories/day energy deficit diet to follow for two weeks.
  Interventions: Behavioral: Caloric restriction

INTERVENTIONS:
Behavioral: Time restricted feeding — Restrict energy intake window to between 8am and 4pm
  Arms: Time restricted feeding (TRF)
Behavioral: Caloric restriction — Follow a prescribed daily energy deficit of 400 kilocalories without altering nutrient timing
  Arms: Caloric deficit

SUMMARY:
In the modern era, food access is widely available and it is not uncommon for the time between breakfast and a late night snack to exceed 14 hours. The investigators are interested in studying whether limiting this window to 8 hours will have any beneficial effects of human health as has been demonstrated in animal models. Eight men were asked to restrict their energy intake window to between 8 am and 4 pm for two weeks whilst maintaining their habitual diet (quantity and composition). Improvements in skeletal muscle and whole-body insulin sensitivity were observed but these were potentially confounded by an average weight loss of 1 kg. Therefore an additional control group was recruited to follow a daily caloric deficit of ~400 kilocalories without changing the timing of intake.

DETAILED DESCRIPTION:
All participants were monitored for a one week baseline period to establish their habitual physical activity and dietary patterns. This was done using food diaries, interstitial glucose monitors and a combined heart rate + accelerometer device. Participants consumed a standardised evening meal ~12h before visiting the laboratory to assess their metabolic response to a liquid test meal (1g/kg bodyweight dextrose and 0.4g/kg bodyweight protein) using the arterio-venous forearm balance model. Dual-energy X-ray absorptiometry scans, indirect calorimetry measurements and fasted and postprandial vastus lateralis biopsies were also obtained.

From the next day, participants either restricted their daily energy intake window to between 8 am and 4 pm or were prescribed a caloric deficit diet (~400 kilocalories/day) for two weeks. Physical activity, interstitial glucose concentrations and dietary patterns were monitored throughout. After this, participants visited the laboratory again to assess changes in metabolism and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male between 18 and 35 years old
* Body mass index between 18 and 27.5 kg.m^-2
* Regular breakfast consumer, 5 or more days per week
* Moderate physical activity level (PAL between 1.6 and 2)

Exclusion Criteria:

* Smoking
* Any metabolic (e.g. diabetes), endocrine (e.g. hyperthyroidism) or cardiovascular (heart or blood) abnormalities including hypertension.
* Clinically significant abnormalities on screening including ECG abnormalities
* Routine medication that may alter cardiovascular function and blood flow (e.g. blood pressure-lowering drugs or drugs that cause hypertension)
* High alcohol consumption (Routinely >4 units per day)
* Eating attitudes test (EAT-26) score > 20
* On an energy-restricted diet
* Significant body mass fluctuation in previous 3 months (>5%)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in glucose uptake | Pre and post intervention (15 days apart). Fasted blood samples and every 10 min for 3 hours following consumption of carbohydrate + protein drink
  The arterio-venous forearm balance method was used to assess skeletal muscle glucose uptake in micromoles/min.
Change in branched chain amino acid uptake | Pre and post intervention (15 days apart). Fasted blood samples and every 10 min for 3 hours following consumption of carbohydrate + protein drink
  The arterio-venous forearm balance method was used to assess skeletal muscle branched chain amino acid uptake in micromoles/min.
Change in whole-body insulin sensitivity | Pre and post intervention (15 days apart).
  The Matsuda Index was used to calculate an index of whole-body insulin sensitivity using values of fasted and postprandial glucose and insulin. Measured in arbitrary units and higher values indicates increased insulin sensitivity. All individual changes will be reported.

SECONDARY OUTCOMES:
Change in body composition | Pre and post intervention (15 days apart)
  Dual-energy X-ray absorptiometry scans to assess changes in fat mass in kg
Change in body composition | Pre and post intervention (15 days apart)
  Dual-energy X-ray absorptiometry scans to assess changes in fat-free mass in kg
Change in substrate metabolism | Pre and post intervention (15 days apart). In each condition there was one measurement in the fasted state and two measurements in the postprandial state.
  Rates of oxygen consumption and carbon dioxide production were measured using indirect calorimetry. These were used to calculate rates of fat and carbohydrate metabolism in grams/min.

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Tsintzas, PhD, Principal Investigator — University of Nottingham
Locations (1):
- MRC/ARUK Centre for Musculoskeletal Ageing, School of Life Sciences, University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones R, Pabla P, Mallinson J, Nixon A, Taylor T, Bennett A, Tsintzas K. Two weeks of early time-restricted feeding (eTRF) improves skeletal muscle insulin and anabolic sensitivity in healthy men. Am J Clin Nutr. 2020 Oct 1;112(4):1015-1028. doi: 10.1093/ajcn/nqaa192. PMID 32729615